CLINICAL TRIAL: NCT07162597
Title: A Study Evaluating the Effectiveness and Safety of Pulsed Field Ablation Using the FARAPULSE™ System for Electrical Isolation of Pulmonary Veins and Superior Vena Cava
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-426R
Record Dates: First submitted 2025-08-31; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation (Paroxysmal)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pulsed Field Ablation (Experimental): Using the FARAPULSE™ System
  Interventions: Device: Pulsed Field Ablation

INTERVENTIONS:
Device: Pulsed Field Ablation — Pulsed Field Ablation

SUMMARY:
This study is a prospective, single-center, single-arm clinical trial planning to screen and enroll 200 subjects. It aims to evaluate the efficacy and safety of pulsed field ablation (PFA) using the FARAPULSE™ system for pulmonary vein isolation (PVI) and superior vena cava isolation (SVCI) in Chinese patients with paroxysmal atrial fibrillation (PAF). Baseline preoperative data, along with intraoperative and postoperative follow-up information, will be collected. The primary endpoint is the proportion of subjects achieving successful PVI and SVCI using solely the FARAPULSE™ PFA system. Secondary endpoints include long-term procedural success rates and various procedural parameters. Additionally, the incidence of adverse events will be recorded as safety endpoints. The study adopts a single-arm target value design hypothesis, and research data will also be compared with historical data from patients treated with radiofrequency ablation for PVI and SVCI to further evaluate the efficacy of PFA. Subgroup analysis will be conducted in patients with heart failure to assess the efficacy and safety of PFA in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years.
* Documented diagnosis of paroxysmal atrial fibrillation (PAF), defined as typical AF electrographic characteristics (absence of P waves with irregular fibrillatory waves) recorded on 12-lead ECG or symptomatic Holter monitoring, with each episode lasting less than 7 days.
* Symptomatic despite attempted antiarrhythmic drug therapy.
* Scheduled to undergo initial catheter ablation procedure.
* Voluntarily provided written informed consent.

Exclusion Criteria:

* AF secondary to electrolyte imbalance, thyroid disorders, or other reversible/non-cardiac causes.
* Persistent atrial fibrillation.
* Presence of persistent left superior vena cava.
* Contraindications to pulsed field ablation (e.g., left atrial appendage thrombus, post-atrial septal defect device closure, permanent metallic implants in the left atrium) or contraindications to anticoagulant therapy.
* Unsuitable for deep sedation/anesthesia per operator assessment.
* Life expectancy less than 1 year.
* Other conditions deemed inappropriate for inclusion by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
PVI and SVCI | Periprocedural
  The proportion of subjects achieving successful PVI and SVCI using solely the FARAPULSE™ PFA system

SECONDARY OUTCOMES:
Long-term procedural success rates | From the end of the 3-month blanking period post-ablation to the 12-month follow-up
  The percentage of subjects, among the total enrolled, who remained free of recurrence of atrial fibrillation, atrial flutter, or atrial tachycardia, with any episode lasting >10 seconds on standard ECG or >30 seconds on Holter monitoring.
Perioperative complications | From the end of the ablation to the 12-month follow-up
  Serious bradyarrhythmia requiring permanent pacemaker implantation, cardiac tamponade/cardiac perforation, thromboembolic events, severe coronary artery spasm (>90% stenosis), phrenic nerve palsy, acute hemolysis and hemolysis-induced renal failure, vascular access complications requiring surgical or interventional management, atrioesophageal fistula, pulmonary vein stenosis, and death.

OTHER OUTCOMES:
Total procedure time | Periprocedural
  The duration from femoral venous puncture until the removal of all devices from the body
Anesthesia induction time | Periprocedural
  The duration from the administration of anesthetic agents until achieving a satisfactory anesthetic state (allowing initiation of the procedure)
Left atrial operation time | Periprocedural
  The duration from the entry of the ablation catheter into the left atrium until its withdrawal from the left atrium
Right atrial operation time | Periprocedural
  The duration from the withdrawal of the ablation catheter from the left atrium until its complete removal from the body
Number of ablations | Periprocedural
  Total number of ablations, number of ablations for pulmonary vein isolation, and number of ablations for superior vena cava isolation.

IPD SHARING:
Plan to Share IPD: No